CLINICAL TRIAL: NCT05378477
Title: Randomized, Controlled, Assessor-Blinded, Comparative Study to Evaluate Safety & Efficacy of a New Suffocation Product vs an Oligodecene-based Suffocation Product, 1% Permethrin & a Fatty Acids-based Product in Subjects With Head Lice.
Brief Title: A Clinical Trial to Evaluate Efficacy and Safety of a New Suffocating Head Lice Product.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OYS008-0020
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Head Lice; Pediculosis Capitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Test product (Experimental): Hemisqualane & beeswax-based lotion (X92001752), killing lice and nits via suffocation.
  Interventions: Device: X92001752
- RID Super Max Solution (Active Comparator): Oligodecene oil-based lotion, killing lice and nits via suffocation.
  Interventions: Device: RID Super Max Solution
- Nix Crème (Active Comparator): Conventional pesticide, containing 1% permethrin.
  Interventions: Drug: Nix Crème
- Pouxit Végétal (Active Comparator): Fatty acid salt-based lotion, killing lice and nits via suffocation.
  Interventions: Device: Pouxit Végétal

INTERVENTIONS:
Device: X92001752 — The test product is a lotion to be applied on dry hair for 10 minutes and then washed out using shampoo. The product is to be applied on Day 0 and repeated again on Day 7.
  Other Names: Test product
  Arms: Test product
Device: RID Super Max Solution — RID Super Max Solution is a lotion to be applied on dry hair for 10 minutes and then washed out using shampoo. The product is to be applied on Day 0 and repeated again on Day 7.
  Other Names: Reference product 1
  Arms: RID Super Max Solution
Drug: Nix Crème — Nix crème must be applied on dry hair for 10 minutes and then washed out with water. The product is to be applied on Day 0 and repeated again on Day 7.
  Other Names: Reference product 2
  Arms: Nix Crème
Device: Pouxit Végétal — Pouxit Végétal must be applied on dry hair for 30 minutes and then washed out using shampoo. According to the instructions for use, only 1 treatment must be performed.
  Other Names: Reference product 3
  Arms: Pouxit Végétal

SUMMARY:
The present study is set-up to compare in vivo clinical performance and safety of the test product (X92001752) versus 3 other pediculicides (2 medical devices and 1 conventional pesticide).

DETAILED DESCRIPTION:
The present study is set-up to compare in vivo clinical performance and safety of the test product versus a) RID Super Max Solution (oligodecene oil), Nix crème (1% permethrin), and Pouxit Végétal (fatty acid salts). 220 subjects (n=55 per treatment group) with confirmed diagnosis of head lice infestation will be included. To support safety, local and global tolerability, skin and ocular irritation will be assessed and adverse events (AEs) will be registered.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: male / female.
2. Women of childbearing potential is a premenopausal female that is anatomically and physiologically capable of becoming pregnant following menarche.

   Female subjects: are women of childbearing potential who test negative for pregnancy and agree to use a reliable method of birth control or remain abstinent during the study. Methods of contraception considered acceptable include oral contraceptives, contraceptive patch, intrauterine device, vaginal ring, diaphragm with contraceptive gel, or condom with contraceptive gel

   -or are women of non-childbearing potential, defined as: women who have had surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation) or women who are ≥60 years of age.
3. Age: ≥ 12 months of age year of age at the time of enrollment.
4. Subject must have an active head lice infestation defined as at least 5 live lice (adults and/or nymphs) and 5 apparently live nits, present on the scalp and/or hair, as determined by a trained evaluator.
5. Subject is in good general health based on medical history.
6. The subject or his/her parent/legal guardian (from age 12-17), must give written informed consent, after having been oral and written informed about benefits and potential risks of the trial, as well as information regarding the insurance, taken out to cover the subjects participating in the study. A caregiver must sign an informed consent agreement for children not old enough to do so. Children ages 6-11 years of age will be administered a child's assent form. Subject or his/her parent/legal guardian must be capable of understanding and providing written informed consent.
7. Following application and rinsing of the test products, subject agrees not to shampoo, wash, or rinse their hair or scalp until the 24-hour post treatment evaluation has been completed.
8. The subject agrees not to cut or chemically treat their hair while participating in the study.
9. No more than one working male per household may be excluded from evaluation if he is assessed as being lice free by himself or caregiver.
10. Subject agrees to follow all study instructions, including attending all follow-up appointments.
11. Agree to not use any other pediculicides or medicated hair grooming products for the duration of the study (through Day 10 visit).
12. The parent or legal guardian of a child must be willing to have other family members screened for head lice. If other household members are found to have head lice and are eligible, they must be either enrolled in the study OR receive the standard of care at the site and in the same manner as study participants.
13. Have a single place of residence.
14. The subject or his/her parent or legal guardian must give written informed consent, after having been oral and written informed about benefits and potential risks of the trial, as well as details of the insurance taken out to cover the subjects participating in the study.
15. Subjects must agree to not use any other ant-lice treatment for the duration of the study.

Exclusion Criteria:

1. Application of any form of head lice treatment, whether prescription or over-the-counter (OTC), or home remedy for 14 days prior to their screening visit (Visit 1).

Application of any topical medication of any kind on the hair for a period of 48 hours prior to the screening visit.

3. Use of systemic or topical drugs or medications, including systemic antibiotics, which in the opinion of the investigative personnel may interfere with the study results.

4. Known skin allergies, multiple drug allergies or multiple allergies to cosmetic products.

5. History of allergy or hypersensitivity to active ingredients, or constituents of the test products.

6. Subject with any visible skin/scalp condition at the treatment site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test product.

7. Subjects with chronic scalp disorder. 8. Subject or his/her legal guardian who, in the opinion of the investigative personnel, do not understand the subject requirements for study participations and/or may be likely to exhibit poor compliance with the required visits.

9. Females who are pregnant or nursing. 10. Hair longer than mid-back. 11. Subject suspected or known not to follow instructions 12. Previous participation in this study or participation in any other investigational trial within the preceding 14 days.

13. The subject is directly affiliated to the investigator site personnel and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

14. The subject is an Oystershell employee or is an employee of a third-party organizations involved in the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects That Are Lice-free After 2 Treatments With Test Product (Including All Baseline Infestations). | Day 10
  Clinical efficacy is reflected by the % of subjects that are lice-free after 2 topical applications (at day 0 & day 7 respectively) of the test product. In this analysis, all baseline infestations (mild, moderate, severe) have been included. Assessment is performed at study end (visit 4, day 10).
  A mild infestation corresponds to 5-9 lice and/or nymphs A moderate infestation corresponds to 10-24 lice and/or nymphs A severe infestation corresponds to 25 or more lice and/or nymphs

SECONDARY OUTCOMES:
Number of Subjects That Are Lice-free After 2 Treatments With RID Super Max Solution (Including All Baseline Infestations). | Day 10
  Clinical efficacy is reflected by the % of subjects that are lice-free after 2 topical applications (at day 0 & day 7 respectively) of RID Super Max Solution. In this analysis, all baseline infestations (mild, moderate, severe) have been included. Assessment is performed at study end (visit 4, day 10).
  A mild infestation corresponds to 5-9 lice and/or nymphs A moderate infestation corresponds to 10-24 lice and/or nymphs A severe infestation corresponds to 25 or more lice and/or nymphs
Number of Subjects That Are Lice-free After 2 Treatments With Nix crème (Including All Baseline Infestations). | Day 10
  Clinical efficacy is reflected by the % of subjects that are lice-free after 2 topical applications (at day 0 & day 7 respectively) of Nix crème. In this analysis, all baseline infestations (mild, moderate, severe) have been included. Assessment is performed at study end (visit 4, day 10).
  A mild infestation corresponds to 5-9 lice and/or nymphs A moderate infestation corresponds to 10-24 lice and/or nymphs A severe infestation corresponds to 25 or more lice and/or nymphs
Number of Subjects That Are Lice-free After 1 Treatment With Pouxit Végétal (Including All Baseline Infestations). | Day 10
  Clinical efficacy is reflected by the % of subjects that are lice-free after 1 topical applications (at day 0) of Pouxit Végétal. In this analysis, all baseline infestations (mild, moderate, severe) have been included. Assessment is performed at day 7 (last visit).
  A mild infestation corresponds to 5-9 lice and/or nymphs A moderate infestation corresponds to 10-24 lice and/or nymphs A severe infestation corresponds to 25 or more lice and/or nymphs
Effect of All Investigational Treatments on Pruritus (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator. | Day 0, Day 1, Day 7, Day 10
  The occurrence and degree of pruritus is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: the scalp does not itch; Mild: occasional episodes of itching, not bothersome; Moderate: frequent, several times a day, bothersome; Severe: nearly constant, frequent scratching, very bothersome.
Effect of All Investigational Treatments on Scalp Excoriation (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator. | Day 0, Day 1, Day 7, Day 10
  The occurrence and degree of scalp excoriation (breaking of the skin, usually caused by scratching) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no broken skin on the scalp; Mild: one or two areas on the scalp on which skin is broken; Moderate: more than two separate areas of the scalp with broken skin but not generalized across the scalp; Severe: widespread breaking of the skin involving most of the scalp.
Effect of All Investigational Treatments on Paraesthesia (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator. | Day 0, Day 1, Day 7, Day 10
  The occurrence and degree of paraesthesia (tingling or prickling sensation) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no tingling or prickling sensation; Mild: occasional tingling or prickling sensation; Moderate: frequent tingling or prickling sensation; Severe: nearly constant tingling or prickling sensation.
Effect of All Investigational Treatments on Skin Erythema (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator. | Day 0, Day 1, Day 7, Day 10
  The occurrence and degree of skin erythema (redness of the scalp) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no redness of the scalp; Mild: faint, barely perceptible erythema with limited distribution; Moderate: diffuse pink areas of scalp are readily visible; Severe: large areas of the scalp are red.
Effect of All Investigational Treatments on Pyroderma (Local Tolerability Parameter), as Assessed by a Blinded Clinical Investigator. | Day 0, Day 1, Day 7, Day 10
  The occurrence and degree of pyroderma (sores filled with clear fluid, pus or crusting) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no lesions visible on the scalp; Mild: one or two lesions visible with crusting or other evidence of infection; Moderate: presence of more than two lesions with crusting or other evidence of infection, but not generalized across the scalp; Severe: lesions with crusting or other evidence of infection, involving most of the scalp.
Effect of All Investigational Treatments on Eye Irritation, as Assessed by a Blinded Clinical Investigator. | Day 0, Day 1, Day 7, Day 10
  The occurrence and degree of eye irritation (stinging, burning sensation, and/or pain) is rated by the blinded clinical investigator at each visit, using the following scores: none (best outcome), mild, moderate, and severe (worst outcome).
  None: no stinging, burning or pain Mild: slight mild stinging, burning or pain Moderate: moderate stinging, burning or pain Severe: severe stinging, burning or pain.
Global Tolerability, Evaluated at Study End (Visit 4, Day 10) | day 10
  Global tolerability is defined as the general well-being and comfort of the subjects. This parameter is assessed at day 10 in subjects, treated with either test product or reference product, respectively. The subject is asked to score his general feeling at study end and must provide a justification for his/her answer. Scoring was performed as follows: very good (best case), good, moderate, or poor (worst case).
Assessment of Adverse Events Occurring After 1 and/or 2 Treatments With Both Investigational Products. | Study period (10 days) + in case of adverse events: clinical staff will monitor the trial subject's safety from the occurrence of an AE until recovery, return to baseline or a stable state will be achieved.
  Recording Adverse Events and investigating the relationship with the treatment. At each visit (D0: first treatment; D1: 24h post-treatment assessment; D7: second treatment; D10: final assessment), the clinical staff is recording adverse events (if any) and evaluates the correlation with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Susel Gonzalez Acosta, ARNP, Principal Investigator — PI
Locations (1):
- South Fla. Family Health & Research Ctr.LLC, Plantation, Florida, United States

IPD SHARING:
Plan to Share IPD: No